CLINICAL TRIAL: NCT03717636
Title: Prospective and Randomized Comparative Analysis, Between Early or Non-revoked in Day Hospital in Patients With Acute Heart Failure
Brief Title: Early or Non-revoked in Hospital-day in Patients With Acute Heart Failure
Acronym: HospDia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSInCor-ICxHospDia
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Acute Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Independent Medical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital Day (Experimental): Patients in the Hospital-Day group will return for medical evaluation 7-14 days in the specific unit.
  Interventions: Other: medical evaluation
- Outpatient clinic (Other): The patients in control group will return for medical evaluation 30 days at the outpatient clinic.
  Interventions: Other: medical evaluation

INTERVENTIONS:
Other: medical evaluation — return of medical evaluation after discharge

SUMMARY:
Heart failure is one of the major causes of hospitalization in Brazil and worldwide. Recent studies attempt to identify readmission and prognostic markers at the time of discharge from these patients. The reassessment and possibility of early therapeutic adjustment may be relevant in this context. Therefore, the prospective and randomized comparative use of early re-evaluation in Hospital-day versus non-intervention group has not yet been described. The objective of this study was to evaluate the impact on the re-hospitalization rate in 30 days of the early re-evaluation of the patients in the day-hospital versus the non-intervention group in heart failure. For this, a unicentric, randomized and prospective study will be performed, in which the Hospital-Day strategy is performed versus no intervention in a comparative manner. Hospital data (test results, medical outcomes, complications) of patients will be analyzed for safety and effectiveness. The hypothesis of this study is that the Hospital-Day strategy is superior to the non-intervention strategy and causes fewer rehospitalizations within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged> 18 years.
* Presence of decomposed CF III or IV of NYHA characterized by> 1 symptom (dyspnea, orthopnea or edema) + 1 clinical sign (rales, edema, ascites or pulmonary congestion on chest X-ray).
* LVEF <45% on transthoracic echocardiography.
* BNP> 400 pg / mL.
* Clinical condition of hospital discharge.
* Signed consent form.

Exclusion Criteria:

* Pregnancy
* Body mass index greater than 40 kg / m2.
* Chronic obstructive pulmonary disease.
* Acute coronary syndrome.
* Acute myocarditis.
* Valvular heart disease.
* Need to use vasoactive drug.
* Cirrhosis of the liver Child C.
* Chronic dialysis renal insufficiency or creatinine> 3.0 mg / dL.
* Indication of implantation device of artificial stimulation.
* Pulmonary thromboembolism.
* Neoplasm terminal.
* Sepsis or septic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of 30-days rehospitalization rate | 30 days
  30-days rehospitalization rate

SECONDARY OUTCOMES:
Mortality | 30 days
  30-days mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided